CLINICAL TRIAL: NCT05198232
Title: The Effects of Virtual Low-Tempo and High-Tempo Zumba® in Individuals With Developmental Disabilities on Functional Mobility, Aerobic Capacity, Inhibitory Control, Attention, and Balance
Brief Title: The Effects of Virtual Zumba® in Individuals With Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Melissa Pangelinan, Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Virtual Adaptive Zumba
Record Dates: First submitted 2021-11-11; First posted 2022-01-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Developmental Disability; Autism Spectrum Disorder; Down Syndrome; Cerebral Palsy
Keywords: Adaptive Exercise; Virtual Exercise; Executive Functioning; Dance
MeSH Terms: conditions — Developmental Disabilities; Autism Spectrum Disorder; Down Syndrome; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants will be quasi-randomized to one of three groups: control (normal activities), low-tempo Zumba®, and high-tempo Zumba®. This quasi-randomization enables the groups to be matched on relevant demographics (disability type, age, sex). This design will enable the investigators to determine the effects of Zumba® and the impact of exercise tempo.
Who Masked: Participant
Masking Description: The two different tempo groups will participate in the program using separate HIPPA-compliant Zoom sessions in different rooms at the community programs. The high-tempo group will be called Group 1 and the low-tempo group will be called Group 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): This group will complete normal daily activities. The participants will complete pre-test, 10 weeks of normal daily activities, and post-test. No changes to their daily schedule will be made by the researcher, the control group will participate in normal activities as part of their community day program.
- Zumba High Tempo (Experimental): The Zumba high tempo group will complete a 10-week (2x a week; 60 minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®). Each session will consist of: a warm-up (3-5 minutes), 5-6 songs with instruction (40 minutes), and a cool down (5 minutes) for a total of about 60 minutes including rest/water breaks and time to transition. The only difference between the two adapted Zumba® programs will be the speed at which the songs will be played and the number of times through each song. The songs for the high-tempo group will be played at full speed; the songs in the high-tempo group will be repeated to ensure an equal amount of time moving for both groups. All sessions will be video recorded and examined for fidelity. This group will complete pre-test, post-test, and a 4-week follow-up.
  Interventions: Behavioral: Zumba High Tempo
- Zumba Low Tempo (Experimental): The Zumba low tempo group will complete a 10-week (2x a week; 60 minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®). Each session will consist of: a warm-up (3-5 minutes), 5-6 songs with instruction (40 minutes), and a cool down (5 minutes) for a total of about 60 minutes including rest/water breaks and time to transition. The only difference between the two adapted Zumba® programs will be the speed at which the songs will be played and the number of times through each song. The songs for the low-tempo group will be set to three-fourths speed. All sessions will be video recorded and examined for fidelity. This group will complete pre-test, post-test, and a 4-week follow-up.
  Interventions: Behavioral: Zumba Low Tempo

INTERVENTIONS:
Behavioral: Zumba High Tempo — The Zumba high tempo group will complete a 10-week (2x a week; 60 minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®). Each session will consist of: a warm-up (3-5 minutes), 5-6 songs with instruction (40 minutes), and a cool down (5 minutes) for a total of about 60 minutes including rest/water breaks and time to transition. The only difference between the two adapted Zumba® programs will be the speed at which the songs will be played and the number of times through each song. The songs for the high-tempo group will be played at full speed; the songs in the high-tempo group will be repeated to ensure an equal amount of time moving for both groups. All sessions will be video recorded and examined for fidelity. This group will complete pre-test, post-test, and a 4-week follow-up.
  Arms: Zumba High Tempo
Behavioral: Zumba Low Tempo — The Zumba low tempo group will complete a 10-week (2x a week; 60 minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®). Each session will consist of: a warm-up (3-5 minutes), 5-6 songs with instruction (40 minutes), and a cool down (5 minutes) for a total of about 60 minutes including rest/water breaks and time to transition. The only difference between the two adapted Zumba® programs will be the speed at which the songs will be played and the number of times through each song. The songs for the low-tempo group will be set to three-fourths speed. All sessions will be video recorded and examined for fidelity. This group will complete pre-test, post-test, and a 4-week follow-up.
  Arms: Zumba Low Tempo

SUMMARY:
There are critical knowledge gaps that need to be addressed to understand the impact of aerobic exercise programs on relevant functional outcomes in adults with developmental disabilities (DD). This study will build upon previous literature by examining the impact of a 10-week (2x a week; 60-minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®) in adults with DD ages 20-69 (n=58). Participants will be quasi-randomized to one of three groups: control (normal activities), low-tempo Zumba®, and high-tempo Zumba®. The quasi-randomization enables the investigators to ensure similarities in relevant demographic factors (e.g., disability type, age, sex) across the three groups. This design will enable the investigators to determine the effects of Zumba® and the impact of tempo level on relevant outcome measures. Participants will compete testing three times - pre-test, post-test, and a 4-week follow-up test - to determine the immediate and long-term benefits of Zumba®. Changes in functional mobility (Timed Up-And-Go), balance (Clinical Test of Sensory Interaction on Balance), aerobic capacity (6-minute Walk Test), and executive functioning (Flanker) will be assessed. During the program, participants' moderate-to-vigorous physical activity (MVPA) will be measured using accelerometry. Compared to the control group, the investigators hypothesize that both Zumba groups will show an improvement in body composition, balance, functional mobility, executive functioning, aerobic capacity, and MVPA during the program. Moreover, the investigators hypothesize that the high tempo group will improve body composition, balance, functional mobility, executive functioning, aerobic capacity, and MVPA during the program more than the low tempo.

DETAILED DESCRIPTION:
The term developmental disabilities (DD) encompasses a group of long-term disabilities that begin before the age of 18 years and include autism spectrum disorder (ASD), cerebral palsy (CP), Down syndrome (DS), intellectual disabilities (ID), and other similar disabilities. Currently, nearly 17% of children have a DD. Furthermore, the prevalence of DD has grown over the last 8 years; the prevalence of ID and DS has increased by more than 25% (from 2009-2017), and ASD has doubled over this period. Simultaneously, the life expectancy of those with DS has also increased to into the sixties and for those with ID into their seventies creating a growing population of older adults with DD. Despite the increase in life expectancy, individuals with DS and ID do not live as long as typically developing individuals and have a lower quality of life throughout the lifespan. Therefore, interventions are needed to improve the health and quality of life in adults with DD.

Individuals with DD face disproportionate physical health problems. Low cardiorespiratory fitness, low physical activity (PA) levels, poor functional mobility, and greater obesity. Together, these issues lead to secondary health conditions that contribute to early morbidity and reduced quality of life for the growing population of adults with DD. In fact, one study found that two of the leading causes of death for individuals with DD, heart disease and diabetes, were correlated with low levels of PA.

Access to adapted PA and fitness programs may attenuate the risk for health problems, poor quality of life, and early morbidity in this population. Indeed, older adults (>50 years old) with ID with high fitness skills (i.e., cardiorespiratory fitness, grip strength, balance) have much high survival rates over a 5-year period than those with low fitness skills. Indeed, aerobic, strengthening, and combined exercise programs have been found to improve the overall health and well-being of adults (ages 18-75) with ID. Thus, there is a clear need to develop and implement exercise and fitness programs to promote healthy aging and reduce physical health disparities in this underserved population.

Aerobic exercise programs have been found to improve cardiorespiratory fitness, strength, flexibility, mobility, and attention in individuals with DD. However, there are several important limitations that suggest the need for further study. First, many previous studies investigating the efficacy of aerobic programs in individuals with DD did not employ randomized control designs, which reduces the generalizability and increases the bias of study results. If there was a control group, the controls consisted of inactive controls. Rather, the use of active control groups helps to determine how different components of the exercise program (e.g., frequency, intensity, time, or type) impact outcomes. Second, few studies have examined the impact of aerobic exercise programs on functional mobility or balance and attention in adults with DD. These two variables are relevant for the ability to perform activities of daily living independently. Third, few studies have included a retention period to examine the long-term impact of aerobic exercise programs (i.e., beyond the immediate effects of an exercise program) in this population. Lastly, only two studies examined the impact of cognitively-engaging aerobic exercise programs like Zumba® in individuals with DD. Cognitively-engaging aerobic exercise programs may confer a greater impact on cognitive functions like attention compared to typical aerobic exercise programs (e.g., running, cycling, etc.).

Given the limitations of previous studies, there are critical knowledge gaps that need to be addressed to understand the impact of aerobic exercise programs on relevant functional outcomes in adults with developmental disabilities (DD). This study will build upon previous literature by examining the impact of a virtual 10-week (2x a week; 60-minutes per session) adapted aerobic dance intervention (adapted Zumba®) in adults with DD ages 19.04-68.78 (n=57). Participants will be quasi-randomized to one of three groups: control (normal activities), low-tempo Zumba®, and high-tempo Zumba®. The quasi-randomization enables the investigators to ensure similarities in relevant demographic factors (e.g., disability type, age, sex) across the three groups. This design will enable the investigators to determine the effects of Zumba® and the impact of exercise tempo. Participants will compete testing three times - pre-test, post-test, and 4-week follow-up test - to determine the immediate and long-term benefits of Zumba®. Changes in functional mobility (Timed Up-And-Go), balance (Clinical Test of Sensory Interaction on Balance), aerobic capacity (6-minute Walk Test), and executive function (Flanker) will be assessed. During the program, participants' MVPA will be measured using wrist-worn accelerometers.

It is hypothesized that:

1. Compared to controls, both adapted Zumba groups will show an increase in balance, functional mobility, and aerobic capacity (Group x Time Interaction). Follow-up t-tests will reveal a dose-dependent improvement in these outcomes between pre-test and post-test (HT>LT>Controls). Moreover, follow-up t-tests will reveal that the high-tempo group will maintain their improvements 4 weeks after the program (post-test to follow-up), compared to the low-tempo group and control group (HT>LT=Controls).
2. Compared to controls, both adapted Zumba groups will show an increase in EF. Follow-up t-tests will reveal a dose-dependent improvement in EF from pre-test to post-test (HT>LT>Controls). Moreover, follow-up t-tests will reveal that the high-tempo group will maintain their improvements 4 weeks after the program (post-test to follow-up), compared to the low-tempo group and control group (HT>LT=Controls).
3. Compared to controls, both adapted Zumba programs will exhibit greater MVPA levels during the program (Group main effect). A follow-up t-test will reveal a dose-dependent increase in MVPA (HT>LT>Controls).
4. Compared to controls, both adapted Zumba programs will exhibit improvements in body composition (Group x Time interaction). Follow-up t-test will reveal that the high-tempo group will exhibit more improvement compared to the low-tempo group and controls (HT >LT>Controls).

Methods Participants 57 individuals with DD ages 18-60 years will be recruited from three community day programs for adults with DD. Participants will be included if the participants are healthy enough to participate in exercise (based on the Physical Activity Readiness Questionnaire or a physician's letter), 18 years or older, and have a diagnosed DD (e.g., Autism Spectrum Disorder, Down Syndrome, Intellectual Disability, etc.).

Study Design The study will examine the impact of a 10-week (2x a week; 60 minutes per session) virtual adapted aerobic dance intervention (adapted Zumba®) with three groups - control (normal activities), low-tempo Zumba®, and high-tempo Zumba®. This quasi-randomized approach will enable the investigators to match the three groups on relevant demographics (i.e., level of function, age, and diagnosis). This design will enable the investigators to determine the overall effects of Zumba® and the impact of tempo level on outcomes. Participants will compete testing three times - pre-test, post-test, and 4-week post-test - to determine dose-dependent (i.e., tempo) the immediate and long-term benefits of Zumba®.

The adapted Zumba® programs will be administered for 10-week (2x a week; 60 minutes per session) via HIPPA-compliant Zoom. Two certified Zumba® instructors will lead the sessions. Both instructors have experience working with children and adults with DD. The instructors will swap halfway through the program to reduce potential instructor bias in leading the high/low tempo sessions. Each session will consist of: a warm-up (3-5 minutes), 4-5 songs with instruction (40 minutes), and a cool down (5 minutes) for a total of about 60 minutes including rest/water breaks and time to transition. The only difference between the two adapted Zumba® programs will be the tempo at which the songs will be played and the number of times through each song. The songs for the low-tempo group will be set to 3/4-speed. The songs for the high-tempo group will be played at full speed; the songs in the high-tempo group will be repeated to ensure an equal amount of time moving for both groups. All sessions will be video recorded and examined for fidelity. The control group will participate in normal activities as part of their community day program.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy enough to participate in exercise (based on the Physical Activity Readiness Questionnaire or a physician's letter)
* 18 years or older
* have a diagnosed Developmental disability (e.g., Autism Spectrum Disorder, Down Syndrome, Intellectual Disability, etc.).

Exclusion Criteria:

* Did not participate in 50% or more of the sessions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory functioning using the 6-minute Walk Test (6MWT) | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the intervention (for the Zumba groups only)
  The 6MWT is a submaximal exercise test to assess cardiorespiratory functioning. The test includes measures of pre-and post-walk blood pressure, heart rate, blood oxygen levels, and fatigue (Borg Scale). The test consists of walking back and forth between two cones set up at a distance of 15-meters for 6 minutes continuously. The total distance walked in meters is recorded for a single trial. This test is valid for individuals ages 16-80, shows good test-retest reliability (ICC = 0.95), and has been used with adults with DD ages 20-80.
Change in Functional Mobility using the Timed-Up and Go (TUG). | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  TUG is a measure of functional mobility. The test consists of the participant sitting in a chair (with no arms), rising from the chair, walking 3 meters to a cone, turning around, walking back to the chair, and sitting in the chair. The total time to complete each trial is recorded. Participants complete a total of three trials - one practice trial and two formal trials that are averaged. This test is valid for individuals ages 16-70, shows good test-retest reliability (ICC = 0.92), and has been used with adults with DD ages 20-80.
Change in Static Balance using the Biodex Balance SD - modified Clinical Test of Sensory Interaction on Balance. | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post test (for the Zumba groups only)
  The Biodex Balance SD measures the center of pressure while the participant stands on the platform during balance tasks. For the purpose of the present proposal, the modified Clinical Test of Sensory Interaction on Balance will be used. This test has been used with adults with developmental disabilities. For this test, the participant stands barefoot with the feet hip-distance apart. Postural sway is measured during each of four conditions (20 seconds per condition): eyes open standing on a firm surface, eyes closed standing on a firm surface, eyes open standing on a foam surface, and eyes closed standing on a foam surface. A sway score is computed based on the sway amplitude.
Change in Attention/Inhibition using the NIH Toolbox Flanker Test. | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  The Flanker test is a measure of selective attention and inhibition. It is conducted on an iPad. For each trial, the direction of a central arrow will change such that the central arrow will be either congruent or incongruent with flanking arrows (e.g., < < > < < or < < < < <). The participant will select the direction of the central arrow by touching the corresponding left or right arrow on the iPad below the stimuli. The participant completes 6 practice trials and a total of 20 formal trials. The raw score is converted to an uncorrected standard score (mean = 100, sd = 15). The NIH Toolbox Flanker Test has been normed based on a sample of typically developing children and adults ages 3-85 and has been used with adults with developmental disabilities . The test shows good test-retest reliability (ICC = 0.80).
Change in Physical activity levels | Throughout all 20 intervention days.
  Wrist-worn triaxial accelerometer (ActiGraph GT3X, Pensacola, Florida) will be used to measure physical activity levels (i.e., light, moderate, vigorous, very vigorous physical activity) during each adapted Zumba® session. The wear time validation algorithm is Choi, which automatically classifies "non-wear time" for 90 minutes of consecutive zero/nonzero counts. The Freedson cut-points will be used for scoring PA into the following categories: light (0-2689 counts per 60 second), moderate (2690-6166 counts per 60 second), vigorous (6167-9642 counts per 60 second), and very vigorous (>9643 counts per 60 second). The wear time validation and cut-points have been used to evaluate PA in adults with disabilities ages 23-72.

SECONDARY OUTCOMES:
Change in Body mass index | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Body mass index will be measured using a bioelectrical impedance scale (BIA; DC 430-U, Tanita Corporation. Tokyo, Japan). Participants will step onto the scale barefoot and must be still for about 10 seconds.
Change in Weight | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Weight will be measured using a bioelectrical impedance scale (BIA; DC 430-U, Tanita Corporation. Tokyo, Japan). Participants will step onto the scale barefoot and must be still for about 10 seconds.
Change in Body fat percentage | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Body fat percentage will be measured using a bioelectrical impedance scale (BIA; DC 430-U, Tanita Corporation. Tokyo, Japan). Participants will step onto the scale barefoot and must be still for about 10 seconds.
Change in Body Fat Mass | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Body fat mass will be measured using a bioelectrical impedance scale (BIA; DC 430-U, Tanita Corporation. Tokyo, Japan). Participants will step onto the scale barefoot and must be still for about 10 seconds.
Change in Fat free mass | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Fat free mass will be measured using a bioelectrical impedance scale (BIA; DC 430-U, Tanita Corporation. Tokyo, Japan). Participants will step onto the scale barefoot and must be still for about 10 seconds.
Change in Height | Pre-test 1 week prior to intervention, Post-test 1 week after the intervention, Follow-up 4 weeks after the post-test (for the Zumba groups only)
  Height will be measured using a stadiometer. Participants will step onto the stadiometer barefoot and must be still for about 10 seconds as researchers indicate their height.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Munn, Study Director — Auburn University
Locations (1):
- Auburn University School of Kinesiology, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymous participant data will be available through a request to the principal investigator.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 5 years following publication.
Access Criteria: Data will be shared with researchers with a minimum qualification of a master's degree in a relevant field (e.g., special education, neuroscience, exercise physiology, kinesiology, disability studies, adapted physical education).

REFERENCES:
- [Background] Blaskowitz, M., Scott, P., Randall, L., Zelenko, M., Green, M., McGrady, E…, Lonergan, M. (2020) Closing the gap: Identifying self-reported quality of life differences between youth with and without intellectual and developmental disabilities. Inclusion, 8 (3), 241-254.
- [Background] Blomqvist S, Wester A, Sundelin G, Rehn B. Test-retest reliability, smallest real difference and concurrent validity of six different balance tests on young people with mild to moderate intellectual disability. Physiotherapy. 2012 Dec;98(4):313-9. doi: 10.1016/j.physio.2011.05.006. Epub 2011 Sep 13. PMID 23122437
- [Background] Bouzas S, Martinez-Lemos RI, Ayan C. Effects of exercise on the physical fitness level of adults with intellectual disability: a systematic review. Disabil Rehabil. 2019 Dec;41(26):3118-3140. doi: 10.1080/09638288.2018.1491646. Epub 2018 Oct 9. PMID 30301367
- [Background] Carmeli E, Bachar A, Merrick J. Blood parameters in adults with intellectual disability at rest and after endurance exercise. Res Sports Med. 2009;17(2):95-103. doi: 10.1080/15438620902900260. PMID 19479628
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Cleaver S, Hunter D, Ouellette-Kuntz H. Physical mobility limitations in adults with intellectual disabilities: a systematic review. J Intellect Disabil Res. 2009 Feb;53(2):93-105. doi: 10.1111/j.1365-2788.2008.01137.x. Epub 2008 Dec 2. PMID 19067784
- [Background] Cluphf, D., O'Connor, J., & Vanin, S. (2001). Effects of aerobic dance on the cardiovascular endurance of adults with intellectual disabilities. Adapted Physical Activity Quarterly, 18(1).
- [Background] Coppus AM. People with intellectual disability: what do we know about adulthood and life expectancy? Dev Disabil Res Rev. 2013;18(1):6-16. doi: 10.1002/ddrr.1123. PMID 23949824
- [Background] de Winter CF, Hermans H, Evenhuis HM, Echteld MA. Associations of symptoms of anxiety and depression with diabetes and cardiovascular risk factors in older people with intellectual disability. J Intellect Disabil Res. 2015 Feb;59(2):176-85. doi: 10.1111/jir.12049. Epub 2013 Apr 30. PMID 23627768
- [Background] Enkelaar L, Smulders E, van Schrojenstein Lantman-de Valk H, Weerdesteyn V, Geurts AC. Clinical measures are feasible and sensitive to assess balance and gait capacities in older persons with mild to moderate Intellectual Disabilities. Res Dev Disabil. 2013 Jan;34(1):276-85. doi: 10.1016/j.ridd.2012.08.014. Epub 2012 Sep 15. PMID 22985782
- [Background] Freedson PS, Lyden K, Kozey-Keadle S, Staudenmayer J. Evaluation of artificial neural network algorithms for predicting METs and activity type from accelerometer data: validation on an independent sample. J Appl Physiol (1985). 2011 Dec;111(6):1804-12. doi: 10.1152/japplphysiol.00309.2011. Epub 2011 Sep 1. PMID 21885802
- [Background] Frey GC, Stanish HI, Temple VA. Physical activity of youth with intellectual disability: review and research agenda. Adapt Phys Activ Q. 2008 Apr;25(2):95-117. doi: 10.1123/apaq.25.2.95. PMID 18493087
- [Background] Guerra-Balic M, Oviedo GR, Javierre C, Fortuno J, Barnet-Lopez S, Nino O, Alamo J, Fernhall B. Reliability and validity of the 6-min walk test in adults and seniors with intellectual disabilities. Res Dev Disabil. 2015 Dec;47:144-53. doi: 10.1016/j.ridd.2015.09.011. Epub 2015 Sep 29. PMID 26426514
- [Background] Heller T, Sorensen A. Promoting healthy aging in adults with developmental disabilities. Dev Disabil Res Rev. 2013;18(1):22-30. doi: 10.1002/ddrr.1125. PMID 23949826
- [Background] Hilapo, P. E., Olea, C. V. B., Panara-ag, A. B., Felismino, N. A., Valera, A. J., & Jr, R. R. V. (2006). Developing speed, flexibility and endurance of people with developmental disabilities using Zumba. Journal of Sciences, Technology and Arts Research, 2, 47-51.
- [Background] Hilgenkamp TI, Reis D, van Wijck R, Evenhuis HM. Physical activity levels in older adults with intellectual disabilities are extremely low. Res Dev Disabil. 2012 Mar-Apr;33(2):477-83. doi: 10.1016/j.ridd.2011.10.011. Epub 2011 Nov 24. PMID 22119695
- [Background] Ko, T., Han, G., & Cho, B. (2012). Effect of 24 weeks of physical activity therapy on the low leg muscular strength. Journal of Physical Therapy Science, 24(4), 351-353.
- [Background] Joseph, B. M. (2018). The Effects of an 8-Week Zumba® Program for Adults with Intellectual and Developmental Disabilities. ProQuest Dissertations and Theses. Florida Atlantic University, Ann Arbor. Retrieved from http://spot.lib.auburn.edu/login?url=https://www.proquest.com/dissertations-theses/effects-8-week-zumba-sup-®-program-adults-with/docview/2185679189/se-2?accountid=8421
- [Background] Lai B, Lee E, Wagatsuma M, Frey G, Stanish H, Jung T, Rimmer JH. Research Trends and Recommendations for Physical Activity Interventions Among Children and Youth With Disabilities: A Review of Reviews. Adapt Phys Activ Q. 2020 Apr 1;37(2):211-234. doi: 10.1123/apaq.2019-0081. Epub 2020 Mar 3. PMID 32131052
- [Background] Landes SD, Stevens JD, Turk MA. Cause of death in adults with intellectual disability in the United States. J Intellect Disabil Res. 2021 Jan;65(1):47-59. doi: 10.1111/jir.12790. Epub 2020 Oct 12. PMID 33043518
- [Background] Melville CA, Hamilton S, Hankey CR, Miller S, Boyle S. The prevalence and determinants of obesity in adults with intellectual disabilities. Obes Rev. 2007 May;8(3):223-30. doi: 10.1111/j.1467-789X.2006.00296.x. PMID 17444964
- [Background] Oppewal A, Hilgenkamp TIM. Physical fitness is predictive for 5-year survival in older adults with intellectual disabilities. J Appl Res Intellect Disabil. 2019 Jul;32(4):958-966. doi: 10.1111/jar.12589. Epub 2019 Apr 5. PMID 30950160
- [Background] Oppewal A, Hilgenkamp TI, van Wijck R, Evenhuis HM. Cardiorespiratory fitness in individuals with intellectual disabilities--a review. Res Dev Disabil. 2013 Oct;34(10):3301-16. doi: 10.1016/j.ridd.2013.07.005. Epub 2013 Jul 26. PMID 23892875
- [Background] Ptomey LT, Szabo AN, Willis EA, Gorczyca AM, Greene JL, Danon JC, Donnelly JE. Changes in cognitive function after a 12-week exercise intervention in adults with Down syndrome. Disabil Health J. 2018 Jul;11(3):486-490. doi: 10.1016/j.dhjo.2018.02.003. Epub 2018 Feb 26. PMID 29501470
- [Background] Rimmer JH, Rowland JL, Yamaki K. Obesity and secondary conditions in adolescents with disabilities: addressing the needs of an underserved population. J Adolesc Health. 2007 Sep;41(3):224-9. doi: 10.1016/j.jadohealth.2007.05.005. PMID 17707291
- [Background] Rimmer JH, Chen MD, McCubbin JA, Drum C, Peterson J. Exercise intervention research on persons with disabilities: what we know and where we need to go. Am J Phys Med Rehabil. 2010 Mar;89(3):249-63. doi: 10.1097/PHM.0b013e3181c9fa9d. PMID 20068432
- [Background] Segal M, Eliasziw M, Phillips S, Bandini L, Curtin C, Kral TV, Sherwood NE, Sikich L, Stanish H, Must A. Intellectual disability is associated with increased risk for obesity in a nationally representative sample of U.S. children. Disabil Health J. 2016 Jul;9(3):392-8. doi: 10.1016/j.dhjo.2015.12.003. Epub 2015 Dec 17. PMID 26785808
- [Background] Shumway-Cook A, Horak FB. Assessing the influence of sensory interaction of balance. Suggestion from the field. Phys Ther. 1986 Oct;66(10):1548-50. doi: 10.1093/ptj/66.10.1548. No abstract available. PMID 3763708
- [Background] Son S, Jeon B, Kim H. Effects of a walking exercise program for obese individuals with intellectual disability staying in a residential care facility. J Phys Ther Sci. 2016 Mar;28(3):788-93. doi: 10.1589/jpts.28.788. Epub 2016 Mar 31. PMID 27134359
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Wu CL, Lin JD, Hu J, Yen CF, Yen CT, Chou YL, Wu PH. The effectiveness of healthy physical fitness programs on people with intellectual disabilities living in a disability institution: six-month short-term effect. Res Dev Disabil. 2010 May-Jun;31(3):713-7. doi: 10.1016/j.ridd.2010.01.013. Epub 2010 Feb 20. PMID 20172687
- [Background] Zablotsky B, Black LI, Maenner MJ, Schieve LA, Danielson ML, Bitsko RH, Blumberg SJ, Kogan MD, Boyle CA. Prevalence and Trends of Developmental Disabilities among Children in the United States: 2009-2017. Pediatrics. 2019 Oct;144(4):e20190811. doi: 10.1542/peds.2019-0811. PMID 31558576
- [Background] Zelazo PD, Anderson JE, Richler J, Wallner-Allen K, Beaumont JL, Conway KP, Gershon R, Weintraub S. NIH Toolbox Cognition Battery (CB): validation of executive function measures in adults. J Int Neuropsychol Soc. 2014 Jul;20(6):620-9. doi: 10.1017/S1355617714000472. Epub 2014 Jun 24. PMID 24960301
- [Background] Zur O, Ronen A, Melzer I, Carmeli E. Vestibulo-ocular response and balance control in children and young adults with mild-to-moderate intellectual and developmental disability: a pilot study. Res Dev Disabil. 2013 Jun;34(6):1951-7. doi: 10.1016/j.ridd.2013.03.007. Epub 2013 Apr 11. PMID 23584174